CLINICAL TRIAL: NCT01691053
Title: Phase II Trial to Evaluate the Efficacy and Safety of Spironolactone in Hemodialysis Patients
Brief Title: Mineralocorticoid Receptor Antagonists in End Stage Renal Disease
Acronym: MiREnDa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Clinical Trial Center Wuerzburg (CTCW) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MN0511_1; 2011-003179-12 (EudraCT Number); 01KG1202 (Other Grant/Funding Number: German Ministry of Education and Research)
Record Dates: First submitted 2012-09-19; First posted 2012-09-24 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: End Stage Renal Disease / Hemodialysis
Keywords: End stage renal disease; Hemodialysis; Spironolactone; Left ventricular hypertrophy
MeSH Terms: conditions — Kidney Failure, Chronic; Hypertrophy, Left Ventricular | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spironolactone (Active Comparator)
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — 50mg once daily
  Arms: Spironolactone
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
End stage renal disease (ESRD) patients exhibit an extraordinarily high annual mortality. Cardiovascular (CV) causes account for almost half of all-cause mortality. Increased left ventricular mass (LVM) is a common finding in ESRD patients on dialysis and is an independent predictor of survival. Yet, to date there is no established medical treatment to reduce CV morbidity and mortality in ESRD patients on hemodialysis. Blockade of aldosterone action by means of mineralocorticoid receptor antagonists (MRA) provides cardioprotection and improves outcome in heart failure patients. Furthermore, the MRA spironolactone has recently been shown to reduce LVM in patients with mild-to-moderate chronic kidney disease (CKD). The investigators here hypothesize that spironolactone treatment is cardioprotective by reducing LVM in ESRD patients on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Hemodialysis treatment for at least 3 months
* At least 3 dialysis sessions per week
* Written informed consent

Exclusion Criteria:

* Contraindications for cardiac magnet resonance imaging (CMR)
* Mineralocorticoid receptor antagonist treatment within the last 6 months
* Estimated life expectancy < 12 months as judged by the nephrologist
* History of hyperkalemia, defined as pre-dialysis potassium > 6.5 mmol/l occurring ≥ 3 times within the last 3 months prior to enrolment.
* High risk to develop hyperkalemia defined as pre-dialysis potassium > 6.0 mmol/l
* Hypotension (systolic blood pressure < 100 mmHg)
* Planned kidney transplantation (living donor) within the prospected study duration
* Any acute illness within the last 4 weeks precluding a study participation as judged by the nephrologist
* Non-amenorrheic women with child bearing potential without reliable contraception, pregnancy/lactation
* Allergy/hypersensitivity to spironolactone
* Non-compliance suspected or demonstrated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2012-12; Primary Completion 2017-02-14 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Left Ventricular Mass Index | 9 months
  as assessed by cardiac MRI

SECONDARY OUTCOMES:
Cardiac function parameters | 9 months
  cardiac volumes, systolic and diastolic function, cardiac output as measured by cardiac MRI and echocardiography
Office and 24h blood pressure | 9 months
Clinical measures of heart failure severity | 9 months
  New York Heart Association (NYHA) functional class, 6 minute walk test
Vascular function | 9 months
  Carotid intima meda thickness, pulse wave analysis, carotid artery distensibility, flow mediated dilatation of the brachial artery
Biomarkers of heart failure, inflammation and fibrosis | 9 months
Quality of Life - Hospital Anxiety and Depression Scale (HADS) | 9 months
  Quality of life will be measured by analyzing HADS
Cardiac death and/or hospitalization for heart failure | 9 months
Safety measures | 9 months
  Pre-dialysis potassium levels, frequency of hyperkalemic episodes (K>6.5mmol/l), measurement of residual kidney function (if applicable)
Quality of Life - Kidney Disease Quality of Life Instrument (KDQOL-SF36) | 9 months
  Quality of life will be measured by analyzing KDQOL-SF36

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Wanner, MD, Principal Investigator — University Hospital Wuerzburg; Fabian Hammer, MD, PhD, Principal Investigator — University Hospital Wuerzburg; Vera Krane, MD, Principal Investigator — University Hospital Wuerzburg
Locations (3):
- Germany (3):
  - University Hospital Erlangen-Nürnberg, Erlangen
  - University Hospital Frankfurt, Frankfurt
  - University Hospital Wuerzburg, Würzburg

REFERENCES:
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138
- [Derived] Hauser T, Dornberger V, Malzahn U, Grebe SJ, Liu D, Stork S, Nauck M, Friedrich N, Dorr M, Wanner C, Krane V, Hammer F; MiREnDa Study Group; Collaborating investigators (sites). The effect of spironolactone on diastolic function in haemodialysis patients. Int J Cardiovasc Imaging. 2021 Jun;37(6):1927-1936. doi: 10.1007/s10554-021-02176-5. Epub 2021 Feb 5. PMID 33544240
- [Derived] Grebe SJ, Malzahn U, Donhauser J, Liu D, Wanner C, Krane V, Hammer F. Quantification of left ventricular mass by echocardiography compared to cardiac magnet resonance imaging in hemodialysis patients. Cardiovasc Ultrasound. 2020 Sep 16;18(1):39. doi: 10.1186/s12947-020-00217-y. PMID 32938484
- [Derived] Hammer F, Krane V, Stork S, Roser C, Hofmann K, Pollak N, Allolio B, Wanner C. Rationale and design of the Mineralocorticoid Receptor Antagonists in End-Stage Renal Disease Study (MiREnDa). Nephrol Dial Transplant. 2014 Feb;29(2):400-5. doi: 10.1093/ndt/gft409. Epub 2013 Oct 28. PMID 24166468